CLINICAL TRIAL: NCT00317291
Title: Acu/Moxa for Peripheral Neuropathy in Persons With HIV
Brief Title: Acupuncture/Moxibustion for Peripheral Neuropathy in HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT003092 (NIH); AAAB4122
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2009-09

CONDITIONS: Peripheral Neuropathies; HIV Infections
Keywords: Acupuncture; HIV; AIDS; Symptom management; Non-invasive; Complementary Therapies; Treatment Experienced
MeSH Terms: conditions — Peripheral Nervous System Diseases; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Acupuncture Therapy; Moxibustion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture/Moxibustion (Experimental): Acupuncture/Moxibustion for Peripheral Neuropathy in HIV
  Interventions: Procedure: Acupuncture/Moxibustion
- Sham acupuncture/Placebo moxibustion (Sham Comparator): Sham acupuncture/Placebo moxibustion for Peripheral Neuropathy in HIV
  Interventions: Other: Sham acupuncture/Placebo moxibustion

INTERVENTIONS:
Procedure: Acupuncture/Moxibustion — Acupuncture/Moxibustion: 16 scheduled sessions
  Arms: Acupuncture/Moxibustion
Other: Sham acupuncture/Placebo moxibustion — Sham acupuncture/Placebo moxibustion: 16 scheduled sessions
  Arms: Sham acupuncture/Placebo moxibustion

SUMMARY:
This is a sample-size-limited, randomized, blinded (subject and evaluator), sham acupuncture/placebo moxibustion (sham acu/placebo moxa) controlled clinical trial. The subjects in this study will be 50 men and women with HIV infection who have a diagnosis of distal symmetric peripheral neuropathy (DSP). Subjects will be randomized to one of two experimental intervention conditions:

* Condition 1: subjects receive acu/moxa treatment; and
* Condition 2 (Control Group): subjects receive sham acu/placebo moxa.

All subjects in Conditions 1 and 2 will attend 16 scheduled sessions over 15 weeks, be administered the same instruments, and submit their daily symptom diaries for analysis. There will be six weeks of twice weekly treatment sessions, and three follow-up sessions at weeks 9, 11, and 15. All conditions will be identical in duration and be administered by licensed acupuncturists trained in traditional Chinese medicine (TCM).

DETAILED DESCRIPTION:
Subjects in this early-phase clinical trial will be 50 men and women with HIV infection who have a diagnosis of Distal Symmetric Peripheral neuropathy (DSP). This study is a prospective, randomized, sham/placebo controlled, blinded (subject and evaluator), parallel groups clinical trial. Subjects will be randomized to one of two experimental intervention conditions:

* Condition 1: subjects receive Acu/Moxa Treatment; and
* Condition 2 (Control Group): subjects receive Sham acupuncture/Placebo moxibustion (Sham Acu/Placebo Moxa).

Subjects in Conditions 1 and 2 will attend 16 scheduled sessions over 15 weeks. All subjects will: be blinded/masked to treatment assignments, attend the same number of protocol sessions, be administered the same instruments, and submit their symptom diaries for data entry and analysis. After a screening/intake session, randomization and treatment sessions will follow. There will be six weeks of twice weekly treatment sessions, and three follow-up sessions at weeks 9, 11 and 15. All conditions will be identical in duration and be administered by licensed acupuncturists trained in Traditional Chinese Medicine. The aims of this study include:

1. To establish the feasibility of the combined Acupuncture/Moxibustion treatment for 6 weeks of twice weekly sessions, in order to reduce the pain related to DSP among persons with HIV/AIDS, and to estimate the effect size of the Acu/Moxa treatment for a future clinical study. Inclusion of 2-, 4-, and 8-week no-treatment follow-up sessions will establish the maintainability of benefit.
2. To determine the effect of combined Acupuncture/Moxibustion treatment for 6 weeks of twice weekly sessions on reducing symptoms of DSP (aching or burning pain, "pins and needles" sensation, and numbness) among persons with HIV/AIDS.
3. To determine the effect of the combined Acupuncture/Moxibustion treatment for 6 weeks of twice weekly sessions on patient-perceived DSP symptom improvement and quality of life.
4. To evaluate the logistics of a CAM clinical trial on persons with HIV/AIDS experiencing DSP.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are HIV positive or Centers for Disease Control (CDC)-defined AIDS diagnosed subjects who are 18 years of age or older, and have a history of distal symmetrical peripheral neuropathy of the lower extremities (legs and feet) for two months or greater.
* Patients experiencing moderate pain severity.
* Verification from primary provider of subject's: HIV status, diagnosis of DSP, and agreement that patient is clinically suitable for the study.
* Individuals able to successfully complete a mini-mental status exam.
* Individuals who understand and agree to complete daily symptom diaries for the duration of the study.
* Individuals taking antiretroviral combinations must have completed an initial 8 weeks of a stable regime (same drug[s], dose, and frequency) prior to entry into the study.
* Individuals taking chronic pain medications must be on a stable regime (same drug, dose, and frequency) for at least twenty-one (21) days prior to entry into the study.
* Individuals on all other medications which may have neuropathy listed as a side effect must be on a stable regime (same drug[s], dose, and frequency) for at least 21 days prior to entry in the study.

Exclusion Criteria:

* Individuals with an acute medical condition, i.e. pneumocystis carinii pneumonia, tuberculosis, and/or other opportunistic infections or conditions that would require medical attention.
* Individuals with diagnosis of diabetes mellitus, B-12 deficiency
* Topically applied medications to the lower extremities.
* Individuals with alcohol and/or substance dependence.
* Individuals with bleeding tendency
* Currently receiving treatment with corticosteroids
* Use of isoniazid (INH), dapsone, or metronidazole within 8 weeks prior to enrollment.
* Severe heart disease, uncontrolled high blood pressure, lung disease, or renal failure.
* Pregnant women
* Individuals receiving acupuncture currently and less than 6 months prior to enrollment.
* Individuals with a history of receiving moxibustion.
* Individuals currently receiving other types of complementary therapies such as herbs, massage, reiki, etc.
* Individuals with plans for travel, lifestyle change, or other activity that would preclude attending all of the planned study sessions and/or recording daily diary information.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Symptom diary
Gracely Pain Scale

SECONDARY OUTCOMES:
Subjective Peripheral Neuropathy Scale
Clinical Global Impression Scale
Neurological Assessment Form

CONTACTS AND LOCATIONS:
Overall Officials: Joyce K Anastasi, PhD, DrNP, Principal Investigator — Columbia University
Locations (1):
- Columbia University School of Nursing, Acupuncture Laboratory, New York, New York, United States